CLINICAL TRIAL: NCT00527670
Title: Pilot Study to Identify the Influence of Genetic Profile Aberrations on Patients With Recurrent Hernias
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: MO-1057938
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Pathological Processes
Keywords: Genomics
MeSH Terms: conditions — Pathologic Processes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Controls: Healthy patients undergoing laparoscopic surgery for cholelithiasis, appendicitis, and adrenalectomy.
  Interventions: Procedure: Normal Controls
- Recurrent Hernia: Patients presenting for laparoscopic repair of ventral or incisional hernias.
  Interventions: Procedure: Recurrent Hernia

INTERVENTIONS:
Procedure: Normal Controls — The control group will have small slivers of tissue removed from the skin and abdomen during surgery to compare genomic information.
  Groups: Normal Controls
Procedure: Recurrent Hernia — This group will have small slivers of tissue removed from the skin and abdomen during hernia repair surgery to find genetic proof of hernias being inherited.
  Groups: Recurrent Hernia

SUMMARY:
The aim of this study is to compare collagen composition in the skin and fascia of patients with recurrent or incisional hernias versus normal controls. We will identify potential genes responsible for genetic alterations in collagen deposition by using gene chip analysis of the tissue obtained and comparing the hernia group versus controls. The ultimate goal of this study is to identify target genes which may help us eventually predict which patients are at risk for developing post-operative hernias.

DETAILED DESCRIPTION:
This is a prospective, case control pilot study with the aim of identifying potential genetic influences on recurrent hernia formation. Patients with recurrent abdominal hernias will be compared with normal control subjects. The study endpoints will compare tissue collagen I/III ratios between the groups. It will also use gene chip technology to identify potential differences in gene expression between the two groups, followed by confirmation of the differential expression using RT-PCR.

Patients will be enrolled from the surgical clinic population. If they consent to the study, both the hernia group and the control group will have 0.5 x 0.5 x 0.1 cm3 pieces of skin and fascia collected at the time of their surgery. A small piece of tissue will be used for immunofluorescene to study collagen I/III ratios. RNA will be extracted from the rest of the tissue for the genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Hernia Group: Diagnosis of ventral or incisional hernia.
* Control Group: appendicitis, symptomatic cholelithiasis or cholecystitis, adrenal disease necessitating adrenalectomy.
* Scheduled for an appropriate laparoscopic repair of above diagnosis.
* Females only: Not pregnant.

Exclusion Criteria:

* Steroid use
* Severe COPD or pulmonary disorders
* History of a connective tissue disorder
* Presentation for surgery with a diagnosis other than those listed above in inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients at the University of Missouri Healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ramshaw, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No